CLINICAL TRIAL: NCT05001659
Title: The Comparison of the Two Simulators for ACLS Straining:Does the Computer Simulator Have the Same Effectiveness as the Mannequin Simulato
Brief Title: The Comparison of the Two Simulators for ACLS Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Guolin Wang, professor, Tianjin Medical University General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GWang
Record Dates: First submitted 2021-06-23; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Computer Simulator and Mannequin Simulator

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer simulator (Other): training students ACLS by one computer simulator
  Interventions: Other: computer simulator and mannequin simulator
- mannequin simulator (Other): training students ACLS by one mannequin simulator
  Interventions: Other: computer simulator and mannequin simulator

INTERVENTIONS:
Other: computer simulator and mannequin simulator — compared two different training simulators with respect to training effectiveness in ACLS training.

SUMMARY:
Compared two different training simulators(the computer screen-based simulator versus the full-scale mannequin-based simulator) with respect to training effectiveness in ACLS training.At the same time,evaluate the effectiveness of combination of these two simulators(screen-based simulation followed by mannequin-based simulation),so that to find out a new simulation format for ACLS training.

DETAILED DESCRIPTION:
A prospective,single-blinded,randomized controlled study was used.30 first-year residents were randomized to Computer screen-based simulator group(C group),full scale Mannequin-based group(M group) and screen+Mannequin combing group(SM group).After a 30min ACLS lecture and 30min integrated CPR hands-on training,all groups received a pretest.The C group was exposed to two ACLS computer scenarions,M group was exposed to two ACLS mannequin scenario.Each scenario took 10min and followed by 20min debriefing with simulation educator.After the training session,each participant completed by modified'megacode'checklist.

ELIGIBILITY:
Inclusion Criteria:

- training doctors,intern Exclusion Criteria:Standardized training of doctors，Medical students

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
the effection of the two different simulators for ACLS training. | six months
  If all the groups have improvement in konwledge,ACLS and non-technical skills.Compared with C group,M group，the scores of each group were compared

CONTACTS AND LOCATIONS:
Locations (1):
- the Computer Simulator,the Mannequin Simulator, Tianjin, Tianjin Municipality, China